CLINICAL TRIAL: NCT00406354
Title: A Randomized, Double-Blind Comparison of Atomoxetine Versus Placebo in Children and Adolescents With Attention-Deficit/Hyperactivity Disorder and Comorbid Oppositional Defiant Disorder
Brief Title: Comparison of Atomoxetine Versus Placebo in Children and Adolescents With ADHD and Comorbid ODD in Germany
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11149; B4Z-SB-LYDW (Other: Eli Lilly and Company)
Record Dates: First submitted 2006-11-29; First posted 2006-12-04 (Estimated); Results first posted 2010-02-12 (Estimated); Last update posted 2010-02-26 (Estimated); Status verified 2010-02

CONDITIONS: Attention Deficit Hyperactivity Disorder; Oppositional Defiant Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Oppositional Defiant Disorder | interventions — Atomoxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Atomoxetine Fast Titration (Experimental): 0.5 milligram per kilogram (mg/kg) daily dose taken orally for 1 week, then 1.2 mg/kg daily dose taken orally for 8 weeks
  Interventions: Drug: Atomoxetine
- Atomoxetine Slow Titration (Experimental): 0.5 mg/kg daily dose taken orally for 1 week, then 0.8 mg/kg daily dose taken orally for 1 week, then 1.2 mg/kg daily dose taken orally for 7 weeks
  Interventions: Drug: Atomoxetine
- Placebo (Placebo Comparator): matching placebo daily dose taken orally
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Atomoxetine — Dosage form for the atomoxetine fast and slow titration arms consists of 2.5 mg, 10 mg, 20 mg, 25 mg, and 40 mg capsules. Double-blind treatment will consist of 3 capsules taken once per day for approximately 9 weeks.
  Other Names: LY139603; Strattera
  Arms: Atomoxetine Fast Titration; Atomoxetine Slow Titration
Drug: Placebo — Double-blind treatment will consist of 3 matching placebo capsules taken once per day by mouth for approximately 9 weeks.
  Arms: Placebo

SUMMARY:
A three-arm, randomized, double-blind, placebo-controlled, Phase 4, multicenter study to compare the efficacy and safety of atomoxetine versus placebo in children and adolescents aged 6 through 17 years with attention-deficit/hyperactivity disorder (ADHD) and comorbid oppositional defiant disorder (ODD) who are treated as outpatients in Germany. After an initial 3- to 28-day screening and washout phase, participants will be assigned to double-blind treatment with atomoxetine or placebo. A 2 week up-titration period will be succeeded by a 7 week treatment period at the target dose. The primary efficacy measure will be the Swanson, Nolan and Pelham Rating Scale Revised (SNAP-IV) ODD subscale score.

ELIGIBILITY:
Inclusion Criteria:

* Male or female outpatients who are at least 6 years of age, and who will not have reached their 18th birthday
* Diagnosis of ADHD and presence of Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) criteria A through C for ODD (NOTE: diagnosis for conduct disorder not exclusionary)
* Normal intelligence
* Able to swallow capsules

Exclusion Criteria:

* Weigh less than 20 kilogram (kg) or more than 90 kg at study entry
* Prior treatment with atomoxetine
* History of seizure disorder, suicidal risk, alcohol or drug abuse within the past 3 months
* History of severe allergies or multiple adverse drug reactions
* Cardiovascular disorders: hypertension, unexplained cardiac signs or symptoms, QT (measure of the time between the start of the Q wave and the end of the T wave in the heart's electrical cycle) prolongation , inherited cardiac disorders

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 181 (Actual)
Dates: Start 2006-11; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (6):
- Germany (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Berlin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Düsseldorf
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fulda
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hamburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Heppenheim an der Bergstrasse
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., München

REFERENCES:
- [Derived] Bangs ME, Wietecha LA, Wang S, Buchanan AS, Kelsey DK. Meta-analysis of suicide-related behavior or ideation in child, adolescent, and adult patients treated with atomoxetine. J Child Adolesc Psychopharmacol. 2014 Oct;24(8):426-34. doi: 10.1089/cap.2014.0005. Epub 2014 Jul 14. PMID 25019647
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Period: All Randomized Patients
Arm/Group | Atomoxetine Fast Titration | Atomoxetine Slow Titration | Placebo
Started | 60 | 61 | 60
Completed | 60 | 61 | 59 (One patient was randomized but never received study treatment.)
Not Completed | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 1
Period: All Randomized and Treated Patients
Arm/Group | Atomoxetine Fast Titration | Atomoxetine Slow Titration | Placebo
Started | 60 | 61 | 59
Completed | 44 | 48 | 37
Not Completed | 16 | 13 | 22
Not completed — Lack of Efficacy | 7 | 4 | 17
Not completed — Adverse Event | 6 | 2 | 1
Not completed — Parent/Caregiver Decision | 2 | 6 | 1
Not completed — Withdrawal by Subject | 1 | 1 | 2
Not completed — Physician Decision | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Atomoxetine Fast Titration | Atomoxetine Slow Titration | Placebo | Total
Number analyzed (Participants) | 60 | 61 | 59 | 180
Age Continuous [Mean (Standard Deviation); unit: years] | 11.1 (2.88) | 10.8 (3.39) | 11.1 (2.77) | 11.0 (3.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 11 | 28
  Male | 51 | 53 | 48 | 152
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 60 | 60 | 58 | 178
  African | 0 | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  Germany | 60 | 61 | 59 | 180
Prior Therapy: Attention-Deficit/Hyperactive Disorder (ADHD), Oppositional Defiant Disorder (ODD) [Number; unit: participants] — Summarizes number of participants who received previous attention-deficit/hyperactive disorder (ADHD) and/or oppositional defiant disorder (ODD) therapy, by medication and non-medication categories. NOTE: Because some participants may have received one or more types of ADHD and/or ODD therapies while others may not, the breakdown of prior therapies by treatment group does not equal the number of participants in each treatment group.
  participants
    Previous treatment with stimulants | 23 | 28 | 29 | 80
    Previous psychotropic medication | 3 | 0 | 3 | 6
    Previous non-drug treatment | 6 | 9 | 9 | 24
    Previous psychotherapy | 8 | 7 | 5 | 20
Summary of ADHD Diagnosis [Number; unit: participants] — Breakdown of ADHD diagnosis in accordance with the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV).
  participants
    ADHD - combined type | 44 | 45 | 47 | 136
    ADHD - predominantly inattentive type | 13 | 14 | 8 | 35
    ADHD - predominantly hyperactive-impulsive type | 3 | 2 | 4 | 9
Summary of ODD Diagnosis [Number; unit: participants] — Breakdown of ODD diagnosis in accordance with the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV).
  participants
    Conduct disorder | 14 | 16 | 14 | 44
    Oppositional defiant disorder | 44 | 45 | 45 | 134
    Disruptive behavior disorder not specified | 1 | 0 | 0 | 1
    Adjustment disorder, emotion, conduct disturbance | 1 | 0 | 0 | 1
Clinical Global Impressions - Severity (CGI-S): ADHD Score [Mean (Standard Deviation); unit: units on a scale] — The physician-rated CGI-S ADHD subscale measures the participant's overall severity of ADHD symptoms (1=normal, not at all ill; 7=among the most extremely ill patients) during the last 7 days.
  units on a scale | 5.0 (0.77) | 5.2 (0.79) | 5.1 (0.74) | 5.1 (0.77)
Clinical Global Impressions - Severity (CGI-S): Combined ADHD and ODD Scores [Mean (Standard Deviation); unit: units on a scale] — The physician-rated CGI-S Combined ADHD and ODD subscale measures the participant's overall severity of both ADHD and ODD symptoms (1=normal, not at all ill; 7=among the most extremely ill patients) during the last 7 days.
  units on a scale | 4.9 (0.77) | 5.4 (0.73) | 5.1 (0.71) | 5.1 (0.76)
Clinical Global Impressions - Severity (CGI-S): ODD Score [Mean (Standard Deviation); unit: units on a scale] — The physician-rated CGI-S ODD subscale measures the participant's overall severity of ODD symptoms (1=normal, not at all ill; 7=among the most extremely ill patients) during the last 7 days.
  units on a scale | 4.9 (0.92) | 5.3 (0.83) | 5.0 (0.86) | 5.1 (0.88)
German Revised Children's Quality of Life Questionnaire (KINDL-R): Emotional Well-Being Score [Mean (Standard Deviation); unit: units on a scale] — KINDL-R ("Revidierter KINDer Lebensqualitatsfragebogen, revised version"), a validated German quality of life (QOL) questionnaire, provides parents' views on their child's emotional QOL. It consists of 24 items covering 6 QOL related dimensions (subscales) and 7 additional items assessing chronic illness. Each item is rated on a 5-point scale (1=never; 5=all the time). Lowest possible score for the Emotional Well-Being subscale is 0; the highest possible score is 100. Scores were normalized between 0 and 100, irrespective of the number of items per subscore. Higher scores indicate better QOL.
  units on a scale | 72.9 (18.58) | 72.5 (17.28) | 70.1 (15.92) | 71.9 (17.22)
German Revised Children's Quality of Life Questionnaire (KINDL-R): Family Score [Mean (Standard Deviation); unit: units on a scale] — KINDL-R ("Revidierter KINDer Lebensqualitatsfragebogen, revised version"), a validated German quality of life (QOL) questionnaire, provides parents' views on their child's emotional QOL. It consists of 24 items covering 6 QOL related dimensions (subscales) and 7 additional items assessing chronic illness. Each item is rated on a 5-point scale (1=never; 5=all the time). The lowest possible score on the Family subscale is 0; the highest possible score is 100. Scores were normalized between 0 and 100, irrespective of the number of items per subscore. Higher scores indicate better QOL.
  units on a scale | 58.7 (20.17) | 57.6 (20.73) | 52.3 (20.50) | 56.2 (20.55)
German Revised Children's Quality of Life Questionnaire (KINDL-R): Friends Score [Mean (Standard Deviation); unit: units on a scale] — KINDL-R ("Revidierter KINDer Lebensqualitatsfragebogen, revised version"), a validated German quality of life (QOL) questionnaire, provides parents' views on their child's emotional QOL. It consists of 24 items covering 6 QOL related dimensions (subscales) and 7 additional items assessing chronic illness. Each item is rated on a 5-point scale (1= never; 5= all the time). The lowest possible score on the Friends subscale is 0; the highest possible score is 100. Scores were normalized between 0 and 100, irrespective of the number of items per subscore. Higher scores indicate better QOL.
  units on a scale | 58.2 (21.56) | 53.9 (21.23) | 54.2 (23.34) | 55.4 (22.02)
German Revised Children's Quality of Life Questionnaire (KINDL-R): Physical Well-Being Score [Mean (Standard Deviation); unit: units on a scale] — KINDL-R ("Revidierter KINDer Lebensqualitatsfragebogen, revised version"), a validated German quality of life (QOL) questionnaire, provides parents' views on their child's emotional QOL. It consists of 24 items covering 6 QOL related dimensions (subscales) and 7 additional items assessing chronic illness. Each item is rated on a 5-point scale (1= never; 5= all the time). The lowest possible score on the Physical Well-Being subscale is 0; highest possible score is 100. Scores were normalized between 0 and 100, irrespective of the number of items per subscore. Higher scores indicate better QOL.
  units on a scale | 79.8 (18.53) | 75.9 (19.99) | 81.5 (16.78) | 79.0 (18.54)
German Revised Children's Quality of Life Questionnaire (KINDL-R): School Score [Mean (Standard Deviation); unit: units on a scale] — KINDL-R ("Revidierter KINDer Lebensqualitatsfragebogen, revised version"), a validated German quality of life (QOL) questionnaire, provides parents' views on their child's emotional QOL. It consists of 24 items covering 6 QOL related dimensions (subscales) and 7 additional items assessing chronic illness. Each item is rated on a 5-point scale (1= never; 5= all the time). The lowest possible score on the School subscale is 0; the highest possible score is 100. Scores were normalized between 0 and 100, irrespective of the number of items per subscore. Higher scores indicate better QOL.
  units on a scale | 62.2 (16.74) | 61.5 (20.62) | 62.4 (15.06) | 62.0 (17.50)
German Revised Children's Quality of Life Questionnaire (KINDL-R): Self Esteem Score [Mean (Standard Deviation); unit: units on a scale] — KINDL-R ("Revidierter KINDer Lebensqualitatsfragebogen, revised version"), a validated German quality of life (QOL) questionnaire, provides parents' views on their child's emotional QOL. It consists of 24 items covering 6 QOL related dimensions (subscales) and 7 additional items assessing chronic illness. Each item is rated on a 5-point scale (1= never; 5= all the time). The lowest possible score on the Self Esteem subscale is 0; the highest possible score is 100. Scores were normalized between 0 and 100, irrespective of the number of items per subscore. Higher scores indicate better QOL.
  units on a scale | 55.4 (18.48) | 52.0 (18.71) | 50.4 (18.92) | 52.6 (18.71)
German Revised Children's Quality of Life Questionnaire (KINDL-R): Total Quality of Life Score [Mean (Standard Deviation); unit: units on a scale] — KINDL-R ("Revidierter KINDer Lebensqualitatsfragebogen, revised version"), a validated German quality of life (QOL) questionnaire, provides parents' views on their child's emotional QOL. It consists of 24 items covering 6 QOL related dimensions (subscales) and 7 additional items assessing chronic illness. Each item is rated on a 5-point scale (1= never; 5= all the time). The lowest possible score in the Total QOL score is 0; the highest possible score is 100. Scores were normalized between 0 and 100, irrespective of the number of items per subscore. Higher scores indicate better QOL.
  units on a scale | 64.5 (12.43) | 62.4 (12.92) | 61.8 (13.02) | 62.9 (12.78)
Impact on Family Scale (FaBel): Total Impact Score [Mean (Standard Deviation); unit: units on a scale] — Family burden is assessed by the FaBel questionnaire (German version of the Impact on Family Scale). Questionnaire is answered by participant's caregiver and contains 33 Likert-scaled items to assess general negative impact (of a disability, disorder, disease) on parents, description of social relationships, concern for siblings, financial impact, problems in coping as well as a total score. Each item is rated on a 4-point scale (1=fully applies, 4=applies not at all). Total scores range from 24-96. Higher scores correspond to higher family burden.
  units on a scale | 53.3 (12.88) | 54.1 (13.15) | 53.9 (12.83) | 53.8 (12.89)
Investigator-Rated Individual Target Behaviors (ITB-Inv): Frequency Score [Mean (Standard Deviation); unit: units on a scale] — ITB-Inv assesses frequency and intensity of individually-defined target behaviors. The investigator defines 3 individual behavior problems based on interviews & additional information. Those most impairing for the child or stressful for the parents will be chosen as target behavior. Frequency of each target behavior during the last 7 days is rated on a 6-point scale (0=never to 5=always) with 0 as lowest possible score and 15 the highest possible score.
  units on a scale | 10.9 (2.03) | 11.4 (2.06) | 11.3 (2.67) | 11.2 (2.27)
Investigator-Rated Individual Target Behaviors (ITB-Inv): Intensity Score [Mean (Standard Deviation); unit: units on a scale] — ITB-Inv assesses frequency and intensity of individually-defined target behaviors. The investigator defines 3 individual behavior problems based on interviews & additional information. Those most impairing for the child or stressful for the parents will be chosen as target behavior. Intensity during the last 7 days is rated on a 10-point scale (0=no problems to 9=most severe problems) with the lowest possible score of 0 and the highest possible of 27.
  units on a scale | 21.3 (3.62) | 22.1 (3.39) | 20.5 (3.57) | 21.3 (3.56)
Parent-Rated Attention-Deficit Scale (FBB-HKS): Total Score, Severity [Mean (Standard Deviation); unit: units on a scale] — FBB-HKS ("Fremdbeurteilungsbogen fur Hyperkinetische Storungen"), the German, parent-rated scale for attention-deficit, is a 20-item rating scale which describes ADHD symptom criteria of DSM-IV and is grouped based upon the 3 ADHD domains: inattention (items 1-9); hyperactivity (items 10-16); impulsivity (items 17-20). Parents rated symptom severity of each item during the last 7 days on a 0 to 3 scale (0=not at all to 3=very much). The total score was calculated for ADHD overall (sum of ratings for items 1-20, divided by 20). High scores indicate high severity of symptoms.
  units on a scale | 2.0 (0.62) | 2.0 (0.54) | 1.9 (0.52) | 2.0 (0.56)
Parent-Rated Oppositional Defiant/Conduct Disorders Scale (FBB-SSV): Total Score, Severity [Mean (Standard Deviation); unit: units on a scale] — FBB-SSV ("Fremdbeurteilungsbogen fur Storungen des Sozialverhaltens"), the German, parent-rated oppositional defiant/conduct disorders scale, covers 23 criteria for ODD and 25 for conduct disorder (CD) in four sections. Parents rated symptom severity of each item during the last 7 days on a 0 to 3 scale (0=not at all to 3=very much). The total score was calculated for ODD/CD overall (sum of ratings for items 1-17, divided by 17). Higher scores indicate higher severity of symptoms.
  units on a scale | 1.4 (0.53) | 1.4 (0.49) | 1.4 (0.56) | 1.4 (0.52)
Swanson, Nolan & Pelham Rating Scale - Revised (SNAP-IV): ADHD Inattention Subscale Score [Mean (Standard Deviation); unit: units on a scale] — The SNAP-IV, ADHD Inattention subscale (items 1-9) scores the intensity of each item during the last seven days on a 0 to 3 scale (0=not at all, 1=just a little, 2=pretty much, 3=very much). The lowest possible score is 0; highest is 27.
  units on a scale | 17.7 (5.23) | 18.3 (4.91) | 17.5 (4.94) | 17.9 (5.01)
Swanson, Nolan & Pelham Rating Scale - Revised (SNAP-IV): Hyperactivity/Impulsivity Score [Mean (Standard Deviation); unit: units on a scale] — The SNAP-IV, ADHD Hyperactivity/Impulsivity subscale (items 10-18) scores the intensity of each item during the last seven days on a 0 to 3 scale (0=not at all, 1=just a little, 2=pretty much, 3=very much). The lowest possible score is 0; highest is 27.
  units on a scale | 19.9 (4.98) | 19.7 (4.76) | 18.9 (4.85) | 19.5 (4.85)
Swanson, Nolan & Pelham Rating Scale - Revised (SNAP-IV): ODD Score [Mean (Standard Deviation); unit: units on a scale] — The SNAP-IV, ODD subscale (items 19-26) scores the intensity of each item during the last seven days on a 0 to 3 scale (0=not at all, 1=just a little, 2=pretty much, 3=very much). The lowest possible score is 0; highest is 24.
  units on a scale | 15.5 (4.07) | 15.6 (3.82) | 15.6 (5.13) | 15.5 (4.35)
Swanson, Nolan & Pelham Rating Scale-Revised (SNAP-IV): ADHD Combined Score [Mean (Standard Deviation); unit: units on a scale] — SNAP-IV is a 26-item scale that includes 1 item for each of 18 symptoms in the DSM-IV diagnosis of ADHD and 1 item for each of 8 symptoms in the DSM-IV diagnosis of ODD. Each item is scored on a 0 to 3 scale (0=Not at All, 1=Just a Little, 2=Pretty Much, 3=Very Much). SNAP-IV yields scores in 3 domains: Inattention (items 1-9: subscore range=0-27), Hyperactivity/impulsivity (items 10-18: subscale range=0-27), and Oppositional (items 19-26: subscale range=0-24). SNAP-IV ADHD combined score (inattention + hyperactivity/impulsivity) range=0-54.
  units on a scale | 37.6 (9.70) | 38.0 (8.91) | 36.4 (9.31) | 37.3 (9.28)

OUTCOME MEASURES:

1. Primary Outcome: Swanson, Nolan and Pelham Rating Scale Revised (SNAP-IV) Oppositional Defiant Disorder: (ODD) Score
Description: The SNAP-IV, a 26-item scale, includes 1 item for each of the 18 symptoms contained in the DSM-IV diagnosis of ADHD and 1 item for each of the 8 symptoms contained in the DSM-IV diagnosis of ODD. Each item is scored on a 0 to 3 scale (0=Not at All, 1=Just a Little, 2=Pretty Much, 3=Very Much). The SNAP-IV yields scores in three domains: Inattention (items 1-9: subscore range=0-27), Hyperact-ivity/Impulsivity (items 10-18: subscale range=0-27), and Oppositional (items 19-26: subscale range=0-24). SNAP-IV: ADHD Combined Scale score (inattention + hyperactivity/impulsivity) ranges from 0-54.
Time Frame: 9 weeks
Population: All participants randomized and receiving at least one dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Atomoxetine Fast Titration | Atomoxetine Slow Titration | Placebo
Number analyzed (Participants) | 60 | 61 | 59
units on a scale | 8.6 (0.7) | 9.0 (0.7) | 12.0 (0.7)
Statistical Analysis 1: Comparison: Atomoxetine Fast Titration vs Atomoxetine Slow Titration vs Placebo; Test type: Superiority or Other; p < .001, Mixed Models Analysis — p-value is from comparison of combined atomoxetine fast group plus atomoxetine slow group versus placebo group at Week 9; Mean Difference (Final Values) = -3.2, 95% CI 2-sided [-5.0 to -1.5], Standard Error of Mean 0.9 — Negative values are in favor of the atomoxetine arms

2. Secondary Outcome: Swanson, Nolan & Pelham Rating Scale - Revised (SNAP-IV): ADHD Combined Score
Description: The SNAP-IV: ADHD Combined Subscale for inattention (items 1-9) and hyperactivity/impulsivity (items 11-19) scores the intensity of each item during the last seven days on a 0 to 3 scale (0=not at all, 1=just a little, 2=pretty much, 3=very much). The lowest possible score is 0; highest is 54.
Time Frame: 9 weeks
Population: All participants randomized and receiving at least one dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Atomoxetine Fast Titration | Atomoxetine Slow Titration | Placebo
Number analyzed (Participants) | 60 | 61 | 59
units on a scale | 22.9 (1.5) | 21.3 (1.4) | 29.6 (1.5)
Statistical Analysis 1: Comparison: Atomoxetine Fast Titration vs Atomoxetine Slow Titration vs Placebo; Test type: Superiority or Other; p < .001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -7.4, 95% CI 2-sided [-11.0 to -3.8], Standard Error of Mean 1.8 — Negative values are in favor of the atomoxetine arms

3. Secondary Outcome: Swanson, Nolan & Pelham Rating Scale - Revised (SNAP-IV): ADHD Inattention Score
Description: The SNAP-IV: ADHD Inattention Subscale (items 1-9) scores the intensity of each item during the last seven days on a 0 to 3 scale (0=not at all, 1=just a little, 2=pretty much, 3=very much). The lowest possible score is 0; highest is 27.
Time Frame: 9 weeks
Population: All participants randomized and receiving at least one dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Atomoxetine Fast Titration | Atomoxetine Slow Titration | Placebo
Number analyzed (Participants) | 60 | 61 | 59
units on a scale | 11.1 (0.7) | 10.0 (0.7) | 14.1 (0.7)
Statistical Analysis 1: Comparison: Atomoxetine Fast Titration vs Atomoxetine Slow Titration vs Placebo; Test type: Superiority or Other; p < .001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -3.5, 95% CI 2-sided [-5.3 to -1.8], Standard Error of Mean 0.9 — Negative values are in favor of the atomoxetine arms

4. Secondary Outcome: Swanson, Nolan & Pelham Rating Scale - Revised (SNAP-IV): Hyperactivity/Impulsivity Score
Description: The SNAP-IV: ADHD Hyperactivity/Impulsivity Subscale (items 10-18) scores the intensity of each item during the last seven days on a 0 to 3 scale (0=not at all, 1=just a little, 2=pretty much, 3=very much). The lowest possible score is 0; highest is 27.
Time Frame: 9 weeks
Population: All participants randomized and receiving at least one dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Atomoxetine Fast Titration | Atomoxetine Slow Titration | Placebo
Number analyzed (Participants) | 60 | 61 | 59
units on a scale | 11.5 (0.8) | 11.1 (0.7) | 15.2 (0.8)
Statistical Analysis 1: Comparison: Atomoxetine Fast Titration vs Atomoxetine Slow Titration vs Placebo; Test type: Superiority or Other; p < .001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -3.9, 95% CI 2-sided [-5.8 to -2.0], Standard Error of Mean 1.0 — Negative values are in favor of the atomoxetine arms

5. Secondary Outcome: Parent-Rated Attention-Deficit Scale (FBB-HKS), Total Score: Severity
Description: FBB-HKS ("Fremdbeurteilungsbogen fur Hyperkinetische Storungen"), the German, parent-rated scale for attention-deficit, is a 20-item rating scale which describes ADHD symptom criteria of DSM-IV and is grouped based upon the 3 ADHD domains: inattention (items 1-9); hyperactivity (items 10-16); impulsivity (items 17-20). Parents rated symptom severity of each item during the last 7 days on a 0 to 3 scale (0=not at all to 3=very much). The total score was calculated for ADHD overall (sum of ratings for items 1-20, divided by 20). Higher scores indicate higher severity of symptoms.
Time Frame: 9 weeks
Population: All participants randomized and receiving at least one dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Atomoxetine Fast Titration | Atomoxetine Slow Titration | Placebo
Number analyzed (Participants) | 60 | 61 | 59
units on a scale | 1.2 (0.1) | 1.1 (0.1) | 1.5 (0.1)
Statistical Analysis 1: Comparison: Atomoxetine Fast Titration vs Atomoxetine Slow Titration vs Placebo; Test type: Superiority or Other; p < .001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-0.6 to -0.2], Standard Error of Mean 0.1 — Negative values are in favor of the atomoxetine arms

6. Secondary Outcome: Parent-Rated Oppositional Defiant/Conduct Disorders Scale (FBB-SSV): Total Score, Severity
Description: FBB-SSV ("Fremdbeurteilungsbogen fur Storungen des Sozialverhaltens"), the German, parent-rated oppositional defiant/conduct disorders scale, covers 23 criteria for ODD and 25 for conduct disorder (CD) in four sections. Parents rated symptom severity of each item during the last 7 days on a 0 to 3 scale (0=not at all to 3=very much). The total score was calculated for ODD/CD overall (sum of ratings for items 1-17, divided by 17). Higher scores indicate higher severity of symptoms.
Time Frame: 9 weeks
Population: All participants randomized and receiving at least one dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Atomoxetine Fast Titration | Atomoxetine Slow Titration | Placebo
Number analyzed (Participants) | 60 | 61 | 59
units on a scale | 0.8 (0.1) | 0.8 (0.1) | 1.0 (0.1)
Statistical Analysis 1: Comparison: Atomoxetine Fast Titration vs Atomoxetine Slow Titration vs Placebo; Test type: Superiority or Other; p = 0.006, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-0.4 to -0.1], Standard Error of Mean 0.1 — Negative values are in favor of the atomoxetine arms

7. Secondary Outcome: Investigator-Rated Individual Target Behaviors (ITB-Inv): Intensity Score
Description: ITB-Inv assesses frequency and intensity of individually-defined target behaviors. The investigator defines 3 individual behavior problems based on interviews and additional information. Those most impairing for the child or stressful for the parents will be chosen as target behavior. Intensity during the last 7 days is rated on a 10-point scale (0=no problems to 9=most severe problems) with the lowest possible score of 0 and the highest possible of 27.
Time Frame: 9 weeks
Population: All participants randomized and receiving at least one dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Atomoxetine Fast Titration | Atomoxetine Slow Titration | Placebo
Number analyzed (Participants) | 60 | 61 | 59
units on a scale | 10.8 (1.1) | 11.9 (1.0) | 14.9 (1.1)
Statistical Analysis 1: Comparison: Atomoxetine Fast Titration vs Atomoxetine Slow Titration vs Placebo; Test type: Superiority or Other; p = 0.010, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -3.5, 95% CI 2-sided [-6.2 to -0.9], Standard Error of Mean 1.4 — Negative values are in favor of the atomoxetine arms

8. Secondary Outcome: Investigator-Rated Individual Target Behaviors (ITB-Inv): Frequency Score
Description: ITB-Inv assesses frequency and intensity of individually-defined target behaviors. The investigator defines 3 individual behavior problems based on interviews and additional information. Those most impairing for the child or stressful for the parents will be chosen as target behavior. Frequency of each target behavior during the last 7 days is rated on a 6-point scale (0=never to 5=always) with 0 as lowest possible score and 15 the highest possible score.
Time Frame: 9 weeks
Population: All participants randomized and receiving at least one dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Atomoxetine Fast Titration | Atomoxetine Slow Titration | Placebo
Number analyzed (Participants) | 60 | 61 | 59
units on a scale | 6.0 (0.6) | 6.6 (0.6) | 8.1 (0.6)
Statistical Analysis 1: Comparison: Atomoxetine Fast Titration vs Atomoxetine Slow Titration vs Placebo; Test type: Superiority or Other; p = 0.010, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.8, 95% CI 2-sided [-3.2 to -0.4], Standard Error of Mean 0.7 — Negative values are in favor of the atomoxetine arms

9. Secondary Outcome: Impact on Family Scale (FaBel), Total Impact Score
Description: Family burden is assessed by the FaBel questionnaire (German version of the Impact on Family Scale). Questionnaire is answered by participant's caregiver and contains 33 Likert-scaled items to assess general negative impact (of a disability, disorder, disease) on parents, description of social relationships, concern for siblings, financial impact, problems in coping as well as a total score. Each item is rated on a 4-point scale (1=fully applies, 4=applies not at all). Total scores range from 24-96. Higher scores correspond to higher family burden.
Time Frame: 9 weeks
Population: All participants randomized and receiving at least one dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Atomoxetine Fast Titration | Atomoxetine Slow Titration | Placebo
Number analyzed (Participants) | 60 | 61 | 59
units on a scale | 54.2 (1.4) | 50.6 (1.4) | 53.8 (1.4)
Statistical Analysis 1: Comparison: Atomoxetine Fast Titration vs Atomoxetine Slow Titration vs Placebo; Test type: Superiority or Other; p = 0.406, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.4, 95% CI 2-sided [-4.9 to 2.0], Standard Error of Mean 1.7 — Negative values are in favor of the atomoxetine arms

10. Secondary Outcome: Clinical Global Impressions - Severity (CGI-S): ADHD Score
Description: The physician-rated CGI-S ADHD measures the participant's overall severity of ADHD symptoms (1=normal, not at all ill; 7=among the most extremely ill patients) during the last 7 days.
Time Frame: 9 weeks
Population: All participants randomized and receiving at least one dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Atomoxetine Fast Titration | Atomoxetine Slow Titration | Placebo
Number analyzed (Participants) | 60 | 61 | 59
units on a scale | 3.5 (0.1) | 3.6 (0.1) | 4.3 (0.1)
Statistical Analysis 1: Comparison: Atomoxetine Fast Titration vs Atomoxetine Slow Titration vs Placebo; Test type: Superiority or Other; p < .001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.7, 95% CI 2-sided [-1.1 to -0.4], Standard Error of Mean 0.2 — Negative values are in favor of the atomoxetine arms

11. Secondary Outcome: Clinical Global Impressions - Severity (CGI-S): ODD Score
Description: The physician-rated CGI-S ODD measures the participant's overall severity of ODD symptoms (1=normal, not at all ill; 7=among the most extremely ill patients) during the last 7 days.
Time Frame: 9 weeks
Population: All participants randomized and receiving at least one dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Atomoxetine Fast Titration | Atomoxetine Slow Titration | Placebo
Number analyzed (Participants) | 60 | 61 | 59
units on a scale | 3.6 (0.2) | 3.5 (0.1) | 4.3 (0.2)
Statistical Analysis 1: Comparison: Atomoxetine Fast Titration vs Atomoxetine Slow Titration vs Placebo; Test type: Superiority or Other; p < .001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.8, 95% CI 2-sided [-1.1 to -0.4], Standard Error of Mean 0.2 — Negative values are in favor of the atomoxetine arms

12. Secondary Outcome: Clinical Global Impressions - Severity (CGI-S): Combined ADHD and ODD Scores
Description: The physician-rated CGI-S Combined ADHD and ODD measures the participant's overall severity of both ADHD and ODD symptoms (1=normal, not at all ill; 7=among the most extremely ill patients) during the last 7 days.
Time Frame: 9 weeks
Population: All participants randomized and receiving at least one dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Atomoxetine Fast Titration | Atomoxetine Slow Titration | Placebo
Number analyzed (Participants) | 60 | 61 | 59
units on a scale | 3.7 (0.1) | 3.5 (0.1) | 4.4 (0.1)
Statistical Analysis 1: Comparison: Atomoxetine Fast Titration vs Atomoxetine Slow Titration vs Placebo; Test type: Superiority or Other; p < .001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.8, 95% CI 2-sided [-1.1 to -0.4], Standard Error of Mean 0.2 — Negative values are in favor of the atomoxetine arms

13. Secondary Outcome: German Revised Children's Quality of Life Questionnaire (KINDL-R): Total Quality of Life Score
Description: KINDL-R ("Revidierter KINDer Lebensqualitatsfragebogen, revised version"), a validated German quality of life (QOL) questionnaire, provides parents' views on their child's emotional QOL. It consists of 24 items covering 6 QOL related dimensions (subscales) and 7 additional items assessing chronic illness. Each item is rated on a 5-point scale (1= never; 5= all the time). The lowest possible score in the Total QOL score is 0; the highest possible score is 100. Scores were normalized between 0 and 100, irrespective of the number of items per subscore. Higher score indicates better QOL.
Time Frame: 9 weeks
Population: All participants randomized and receiving at least one dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Atomoxetine Fast Titration | Atomoxetine Slow Titration | Placebo
Number analyzed (Participants) | 60 | 61 | 59
units on a scale | 66.0 (1.8) | 65.6 (1.8) | 60.7 (1.8)
Statistical Analysis 1: Comparison: Atomoxetine Fast Titration vs Atomoxetine Slow Titration vs Placebo; Test type: Superiority or Other; p = 0.021, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 5.0, 95% CI 2-sided [0.8 to 9.3], Standard Error of Mean 2.2 — Positive values are in favor of the atomoxetine arms

14. Secondary Outcome: German Revised Children's Quality of Life Questionnaire (KINDL-R): Physical Well-Being Score
Description: KINDL-R ("Revidierter KINDer Lebensqualitatsfragebogen, revised version"), a validated German quality of life (QOL) questionnaire, provides parents' views on their child's emotional QOL. It consists of 24 items covering 6 QOL related dimensions (subscales) and 7 additional items assessing chronic illness. Each item is rated on a 5-point scale (1= never; 5= all the time). The lowest possible score on the Physical Well-Being subscale is 0; highest possible score is 100. Scores were normalized between 0 and 100, irrespective of the number of items per subscore. Higher scores indicate better QOL.
Time Frame: 9 weeks
Population: All participants randomized and receiving at least one dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Atomoxetine Fast Titration | Atomoxetine Slow Titration | Placebo
Number analyzed (Participants) | 60 | 61 | 59
units on a scale | 69.1 (2.7) | 71.9 (2.6) | 78.1 (2.6)
Statistical Analysis 1: Comparison: Atomoxetine Fast Titration vs Atomoxetine Slow Titration vs Placebo; Test type: Superiority or Other; p = 0.017, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -7.6, 95% CI 2-sided [-13.8 to -1.4], Standard Error of Mean 3.1 — Positive values are in favor of the atomoxetine arms

15. Secondary Outcome: German Revised Children's Quality of Life Questionnaire (KINDL-R): Emotional Well-Being Score
Description: KINDL-R ("Revidierter KINDer Lebensqualitatsfragebogen, revised version"), a validated German quality of life (QOL) questionnaire, provides parents' views on their child's emotional QOL. It consists of 24 items covering 6 QOL related dimensions (subscales) and 7 additional items assessing chronic illness. Each item is rated on a 5-point scale (1= never; 5= all the time).The lowest possible score for the Emotional Well-Being subscale is 0; highest possible score is 100. Scores were normalized between 0 and 100, irrespective of the number of items per subscore. Higher scores indicate better QOL.
Time Frame: 9 weeks
Population: All participants randomized and receiving at least one dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Atomoxetine Fast Titration | Atomoxetine Slow Titration | Placebo
Number analyzed (Participants) | 60 | 61 | 59
units on a scale | 71.8 (2.3) | 73.0 (2.3) | 66.9 (2.3)
Statistical Analysis 1: Comparison: Atomoxetine Fast Titration vs Atomoxetine Slow Titration vs Placebo; Test type: Superiority or Other; p = 0.050, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 5.5, 95% CI 2-sided [-0.0 to 10.9], Standard Error of Mean 2.8 — Positive values are in favor of the atomoxetine arms

16. Secondary Outcome: German Revised Children's Quality of Life Questionnaire (KINDL-R): Self Esteem Score
Description: KINDL-R ("Revidierter KINDer Lebensqualitatsfragebogen, revised version"), a validated German quality of life (QOL) questionnaire, provides parents' views on their child's emotional QOL. It consists of 24 items covering 6 QOL related dimensions (subscales) and 7 additional items assessing chronic illness. Each item is rated on a 5-point scale (1= never; 5= all the time). The lowest possible score on the Self Esteem subscale is 0; the highest possible score is 100. Scores were normalized between 0 and 100, irrespective of the number of items per subscore. Higher scores indicate better QOL.
Time Frame: 9 weeks
Population: All participants randomized and receiving at least one dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Atomoxetine Fast Titration | Atomoxetine Slow Titration | Placebo
Number analyzed (Participants) | 60 | 61 | 59
units on a scale | 60.1 (2.5) | 57.3 (2.4) | 48.0 (2.4)
Statistical Analysis 1: Comparison: Atomoxetine Fast Titration vs Atomoxetine Slow Titration vs Placebo; Test type: Superiority or Other; p < .001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 10.7, 95% CI 2-sided [4.9 to 16.4], Standard Error of Mean 2.9 — Positive values are in favor of the atomoxetine arms

17. Secondary Outcome: German Revised Children's Quality of Life Questionnaire (KINDL-R): Family Score
Description: KINDL-R ("Revidierter KINDer Lebensqualitatsfragebogen, revised version"), a validated German quality of life (QOL) questionnaire, provides parents' views on their child's emotional QOL. It consists of 24 items covering 6 QOL related dimensions (subscales) and 7 additional items assessing chronic illness. Each item is rated on a 5-point scale (1=never; 5=all the time). The lowest possible score on the Family subscale is 0; the highest possible score is 100. Scores were normalized between 0 and 100, irrespective of the number of items per subscore. Higher scores indicate better QOL.
Time Frame: 9 weeks
Population: All participants randomized and receiving at least one dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Atomoxetine Fast Titration | Atomoxetine Slow Titration | Placebo
Number analyzed (Participants) | 60 | 61 | 59
units on a scale | 63.7 (2.8) | 61.9 (2.7) | 54.7 (2.7)
Statistical Analysis 1: Comparison: Atomoxetine Fast Titration vs Atomoxetine Slow Titration vs Placebo; Test type: Superiority or Other; p = 0.015, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 8.1, 95% CI 2-sided [1.6 to 14.6], Standard Error of Mean 3.3 — Positive values are in favor of the atomoxetine arms

18. Secondary Outcome: German Revised Children's Quality of Life Questionnaire (KINDL-R): Friends Score
Description: KINDL-R ("Revidierter KINDer Lebensqualitatsfragebogen, revised version"), a validated German quality of life (QOL) questionnaire, provides parents' views on their child's emotional QOL. It consists of 24 items covering 6 QOL related dimensions (subscales) and 7 additional items assessing chronic illness. Each item is rated on a 5-point scale (1= never; 5= all the time). The lowest possible score on the Friends subscale is 0; the highest possible score is 100. Scores were normalized between 0 and 100, irrespective of the number of items per subscore. Higher scores indicate better QOL.
Time Frame: 9 weeks
Population: All participants randomized and receiving at least one dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Atomoxetine Fast Titration | Atomoxetine Slow Titration | Placebo
Number analyzed (Participants) | 60 | 61 | 59
units on a scale | 67.1 (2.8) | 61.3 (2.8) | 56.2 (2.8)
Statistical Analysis 1: Comparison: Atomoxetine Fast Titration vs Atomoxetine Slow Titration vs Placebo; Test type: Superiority or Other; p = 0.018, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 8.0, 95% CI 2-sided [1.4 to 14.7], Standard Error of Mean 3.4 — Positive results are in favor of the atomoxetine arms

19. Secondary Outcome: German Revised Children's Quality of Life Questionnaire (KINDL-R): School Score
Description: KINDL-R ("Revidierter KINDer Lebensqualitatsfragebogen, revised version"), a validated German quality of life (QOL) questionnaire, provides parents' views on their child's emotional QOL. It consists of 24 items covering 6 QOL related dimensions (subscales) and 7 additional items assessing chronic illness. Each item is rated on a 5-point scale (1= never; 5= all the time). The lowest possible score on the School subscore is 0; the highest possible score is 100. Scores were normalized between 0 and 100, irrespective of the number of items per subscore. Higher scores indicate better QOL.
Time Frame: 9 weeks
Population: All participants randomized and receiving at least one dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Atomoxetine Fast Titration | Atomoxetine Slow Titration | Placebo
Number analyzed (Participants) | 60 | 61 | 59
units on a scale | 63.4 (2.8) | 67.4 (2.8) | 60.5 (2.8)
Statistical Analysis 1: Comparison: Atomoxetine Fast Titration vs Atomoxetine Slow Titration vs Placebo; Test type: Superiority or Other; p = 0.138, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 4.9, 95% CI 2-sided [-1.6 to 11.5], Standard Error of Mean 3.3 — Positive values are in favor of the atomoxetine arms

20. Secondary Outcome: Number of Participants Discontinuing Treatment
Description: Originally, time to treatment discontinuation was analyzed, deeming participants 'censored' if they reached the end of the observation period, were lost to followup, or withdrew informed consent. Because the median was not reached, the number of participants who discontinued (i.e., those who were not censored) is reported here.
Time Frame: 9 weeks
Population: All participants randomized and receiving at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Atomoxetine Fast Titration | Atomoxetine Slow Titration | Placebo
Number analyzed (Participants) | 60 | 61 | 59
participants
  Age <12 Years | 4 | 8 | 15
  Age >=12 Years | 2 | 5 | 4
Statistical Analysis 1: Comparison: Atomoxetine Fast Titration vs Atomoxetine Slow Titration vs Placebo; Test type: Superiority or Other; p = 0.016, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 2.193, 95% CI [1.160 to 4.146]

21. Secondary Outcome: Number of Patients Who Experienced Clinically Relevant Categories of Adverse Events During Initial Three Weeks of Study Treatment
Description: Number of participants who experienced pre-specified categories of clinically relevant adverse events during the initial three-weeks of study treatment. NOTE: this is a subset of the overall adverse events which are reported by participant and event.
Time Frame: 3 weeks
Population: All randomized participants who received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Atomoxetine Fast Titration | Atomoxetine Slow Titration | Placebo
Number analyzed (Participants) | 60 | 61 | 59
participants
  Nausea or related symptoms | 21 | 18 | 5
  Fatigue or related symptoms | 19 | 14 | 6
  Gastrointestinal complaints | 12 | 8 | 2
  Sleep disturbances | 2 | 2 | 1
Statistical Analysis 1: Comparison: Atomoxetine Fast Titration vs Atomoxetine Slow Titration vs Placebo; Test type: Superiority or Other; p = 0.102, Fisher Exact — p-value is from comparison of atomoxetine fast group versus atomoxetine slow group for any clinically relevant categories of adverse events during the initial three weeks of study treatment

22. Secondary Outcome: Number of Patients Who Experienced Clinically Relevant Categories of Adverse Events During Nine-Week Study Treatment Period
Description: Number of participants who experienced pre-specified categories of clinically relevant adverse events during the nine-week study treatment period. NOTE: this is a subset of the overall adverse events which are reported by participant and event.
Time Frame: 9 weeks
Population: All randomized participants who received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Atomoxetine Fast Titration | Atomoxetine Slow Titration | Placebo
Number analyzed (Participants) | 60 | 61 | 59
participants
  Nausea or related symptoms | 25 | 21 | 6
  Fatigue or related symptoms | 20 | 14 | 6
  Gastrointestinal complaints | 14 | 12 | 3
  Sleep disturbances | 4 | 3 | 2
Statistical Analysis 1: Comparison: Atomoxetine Fast Titration vs Atomoxetine Slow Titration vs Placebo; Test type: Superiority or Other; p = 0.101, Fisher Exact — p-value is from comparison of atomoxetine fast group versus atomoxetine slow group for any clinically relevant categories of adverse events during the nine-week study treatment period

ADVERSE EVENTS:
Time Frame: Adverse events reported by participant and event over the complete nine-week study treatment period (NOTE: includes events within clinically relevant categories reported in Outcome Measures #21 [initial three weeks] and #22 [nine-week treatment period]).
Arm/Group | Atomoxetine Fast Titration | Atomoxetine Slow Titration | Placebo
Serious Adverse Events (participants affected / at risk) | 1/60 | 1/61 | 1/59
Other Adverse Events (participants affected / at risk) | 48/60 | 43/61 | 32/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atomoxetine Fast Titration (N=60) | Atomoxetine Slow Titration (N=61) | Placebo (N=59)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atomoxetine Fast Titration (N=60) | Atomoxetine Slow Titration (N=61) | Placebo (N=59)
Vertigo (Ear and labyrinth disorders) | 3 (3) | 0 (0) | 0 (0)
Mydriasis (Eye disorders) | 7 (7) | 5 (5) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 5 (5) | 6 (7) | 3 (4)
Abdominal pain upper (Gastrointestinal disorders) | 8 (9) | 7 (7) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 4 (4) | 3 (3)
Nausea (Gastrointestinal disorders) | 13 (15) | 12 (12) | 3 (3)
Vomiting (Gastrointestinal disorders) | 9 (11) | 11 (12) | 3 (3)
Fatigue (General disorders) | 21 (22) | 13 (14) | 6 (6)
Pyrexia (General disorders) | 5 (6) | 2 (2) | 3 (3)
Nasopharyngitis (Infections and infestations) | 6 (6) | 2 (3) | 3 (3)
Rhinitis (Infections and infestations) | 3 (3) | 1 (1) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 9 (9) | 7 (7) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 4 (4) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 1 (1) | 3 (3)
Headache (Nervous system disorders) | 15 (24) | 9 (10) | 9 (10)
Aggression (Psychiatric disorders) | 2 (2) | 1 (1) | 4 (4)
Sleep disorder (Psychiatric disorders) | 3 (3) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 5 (5) | 3 (3)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days